CLINICAL TRIAL: NCT02894944
Title: Clinical Trial Phase I for Evaluation of Tolerability and Safety of Replication-competent Adenovirus-mediated Double Suicide Gene Therapy in Combination With Chemotherapy for the Locally Advanced Pancreatic Cancer
Brief Title: Clinical Trial Phase I for Theragene in Combination With Chemotherapy for the Locally Advanced Pancreatic Cancer
Acronym: Theragene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: NewGenPharm Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2016-02
Record Dates: First submitted 2016-08-10; First posted 2016-09-09 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Adenovirus; Gene therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Theragene arm (Experimental): Patients who were treated with Theragene®,Ad5-yCD/mutTKSR39rep-ADP and chemotherapy
  Interventions: Biological: Theragene®,Ad5-yCD/mutTKSR39rep-ADP

INTERVENTIONS:
Biological: Theragene®,Ad5-yCD/mutTKSR39rep-ADP — Theragene®,Ad5-yCD/mutTKSR39rep-ADP is Adenovirus-mediated Double Suicide Gene Therapy

SUMMARY:
Pancreatic cancer is associated with an extremely poor prognosis, reflected by a 5-y survival probability of less than 5% when all stages are combined. At present, only approximately 10%-20% of patients are considered candidates for curative resection. The majority of patients (50%-60%) are present with metastatic disease, and substantial number of patients (approximately 30%-40%) are considered ''locally advanced'' at the time of diagnosis.

Replication-competent Adenovirus-mediated Double Suicide Gene Therapy (Theragene®,Ad5-yCD/mutTKSR39rep-ADP) showed an anti-cancer effect in patients with prostatic cancer in phase I study. From the experience of prostatic cancer, the safety of combination with standard chemotherapy with Theragene treatment is assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cancer stage 3
* Patients with histologically confirmed pancreatic adenocarcinoma
* Patients with no evidence of peritoneal or hematogenous metastasis
* Patients with ECOG performance status 0-2
* Patients with renal function (Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min/m²)
* Patients with bone marrow function (WBC > 4,000/uL or absolute neutrophil count ≥ 1500/uL, PLT ≥ 100,000/uL, and Hemoglobin > 10 g/dL)
* Patients with liver function (Bilirubin < 2.0 mg/dL and SGOT and SGPT < 2.5 times upper limit of normal (ULN))
* Patients with agreement with informed consent
* Male patients with contraception

Exclusion Criteria:

* Female patients with childbearing age or pregnancy or breast feeding
* Patients with a history of chemotherapy within 5 years
* Patients with a history of radiation on more than 25% of bone marrow
* Patients with unknown stage or recurrent pancreatic cancer
* Patients with a history of skin cancer except malignant melanoma or malignancy except stage 0 cervical cancer
* Patients with a history of major surgery except laparoscopic exam, endoscopic ultrasound, stenting, or PEG/PEJ placement
* Patients with active or uncontrolled infection
* Patients with immunosuppression or susceptibility to viral infection
* Patients with HIV infection, chronic hepatitis B, chronic hepatitis C, or liver cirrhosis
* Patients with a history of allergy to clinical trial medications
* Patients who are considered as inappropriate candidate by investigators

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v4.03 | 8 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v4.03 | 12 weeks
Tumor response | 8 weeks
Time to disease progression | 6.5 months
Detection of Infected Adenovirus in blood and urine assessed by PCR | 8 weeks
Detection of adenoviral DNA in blood by PCR | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee JC, Shin DW, Park H, Kim J, Youn Y, Kim JH, Kim J, Hwang JH. Tolerability and safety of EUS-injected adenovirus-mediated double-suicide gene therapy with chemotherapy in locally advanced pancreatic cancer: a phase 1 trial. Gastrointest Endosc. 2020 Nov;92(5):1044-1052.e1. doi: 10.1016/j.gie.2020.02.012. Epub 2020 Feb 19. PMID 32084409